CLINICAL TRIAL: NCT02122198
Title: Vascular Mechanisms for the Effects of Loss of Ovarian Hormone Function on Cognition in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 14-0193; UL1TR001082 (NIH)
Record Dates: First submitted 2014-04-22; First posted 2014-04-24 (Estimated); Results first posted 2022-01-10 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Cognitive Impairment; Executive Dysfunction; Endothelial Dysfunction; Cardiovascular Disease
Keywords: Cognitive impairment; Executive function; Arterial stiffness; Endothelial function; Menopause; Women's health; Hormone therapy; functional MRI
MeSH Terms: conditions — Cognitive Dysfunction; Cardiovascular Diseases | interventions — Leuprolide; Estradiol; Medroxyprogesterone; Medroxyprogesterone Acetate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Monthly placebo injections for 6 months under parent study (FAME) protocol (NCT01712230)
  Interventions: Drug: Placebo
- GnRH agonist (Active Comparator): Monthly injections of leuprolide acetate 3.75mg for 9 months; first 6 months under parent study (FAME) protocol (NCT01712230); months 6-9 under sub-study protocol.
  Weekly application of estradiol patch 0.075mg/d months 6-9.
  Daily medroxyprogesterone acetate 5mg by mouth for 12 days at week 30.
  Interventions: Drug: Leuprolide acetate; Drug: Estradiol; Drug: Medroxyprogesterone

INTERVENTIONS:
Drug: Leuprolide acetate — Lupron 3.75 mg for depot suspension delivered by monthly intramuscular injection for 9 months. First 6 months under parent study (FAME) protocol (NCT01712230); months 6-9 under sub-study.
  Other Names: Lupron
  Arms: GnRH agonist
Drug: Estradiol — Climara transdermal patch 0.075mg/day applied weekly months 6-9
  Other Names: Climara
  Arms: GnRH agonist
Drug: Medroxyprogesterone — Provera 5mg tablets once daily by mouth for 12 days beginning at week 30.
  Other Names: Provera
  Arms: GnRH agonist
Drug: Placebo — placebo
  Arms: Placebo

SUMMARY:
Complaints about memory and thinking are common in women as they go through menopause and estrogen levels fall. The ovarian hormone estrogen is important for supporting normal cognitive function, and changes in brain activity and function occur when estrogen levels are decreased. Estrogen is also important for maintaining healthy blood vessels which also support normal cognitive function. In Alzheimer's disease and other types of dementia, there is significant damage to the blood vessels in the brain. This study will test whether changes in brain activity and function with the loss of estrogen are related to changes in vascular function. The investigators will measure vascular function using ultrasound, and brain activity using MRI scans in women who are enrolled in the Females, Aging, Metabolism and Exercise (FAME) study (NCT01712230). In the FAME study, healthy premenopausal women either take a medication to decrease their estrogen levels, or a placebo. This sub-study may provide new information about how estrogen affects vascular function and cognitive function, and lead to new ways to prevent or delay cognitive impairment or dementia.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers will be healthy women aged 40 to 60 years
2. Are enrolled in the parent FAME study (NCT01712230).

The Investigators will consent up to 80 subjects with the aim of enrolling 17 in each of the 2 groups (placebo, GnRH agonist).

Exclusion Criteria:

1. mini-mental state examination (MMSE) score 27 or less
2. history of neurologic disease or major psychiatric illness
3. major depressive episode within the past 12 months
4. history of learning disability
5. less than high-school education
6. current smoking
7. use of psychoactive medications in the past 3 months (stable use of anti- depressant medication is allowed)
8. contraindications to MRI scanning

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy women aged 40 to 60 years.
Enrollment: 17 (Actual)
Dates: Start 2014-09-08 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry L Hildreth, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - University of Colorado Boulder Intermountain Neuroimaging Consortium, Boulder, Colorado

RESULTS

PARTICIPANT FLOW:
Groups:
- GnRH Agonist: Monthly injections of leuprolide acetate 3.75mg for 9 months; first 6 months under parent study (FAME) protocol (NCT01712230); months 6-9 under sub-study protocol.
  Weekly application of estradiol patch 0.075mg/d months 6-9.
  Daily medroxyprogesterone acetate 5mg by mouth for 12 days at week 30.
  Leuprolide acetate: Lupron 3.75 mg for depot suspension delivered by monthly intramuscular injection for 9 months. First 6 months under parent study (FAME) protocol (NCT01712230); months 6-9 under sub-study.
  Estradiol: Climara transdermal patch 0.075mg/day applied weekly months 6-9
  Medroxyprogesterone: Provera 5mg tablets once daily by mouth for 12 days beginning at week 30.
Period: Overall Study
Arm/Group | Placebo | GnRH Agonist
Started | 5 | 12
Completed | 3 | 10
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | GnRH Agonist | Total
Number analyzed (Participants) | 5 | 12 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (2.5) | 47.7 (4.0) | 47.1 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 12 | 17
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 3 | 12 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 3 | 11 | 14
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Changes in Prefrontal Cortex Brain Activation at 6 Months
Description: Changes in patterns of brain activation in the prefrontal cortex using functional magnetic resonance imaging (fMRI) during a task of working memory will be measured at baseline, 6 months, and 9 months (GnRH agonist arm only). Beta weight is the percent signal change on the FMRI from one condition to another. The FMRI is measuring blood oxygen levels and blood flow in different regions of the brain and using that to determine activity changes in the brain. A positive number/increase indicates more blood flow and brain activity in that area.
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: beta-weight
Arm/Group | Placebo | GnRH Agonist
Number analyzed (Participants) | 2 | 7
beta-weight
  Frontal Pole (L) | 90.64 (3.88) | -62.20 (57.61)
  Frontal Orbital Cortex (L) | 28.07 (37.48) | -79.04 (71.85)
  Superior Frontal Gyrus (R) | 92.45 (33.66) | -53.05 (41.13)

2. Primary Outcome: Changes in Prefrontal Cortex Brain Activation at 9 Months
Description: as for outcome 1
Time Frame: Baseline, 9 months
Population: This outcome measure was only collected for a subset of the GnRH Agonist group.
Measure: Mean (Standard Deviation); unit: beta-weight
Arm/Group | GnRH Agonist
Number analyzed (Participants) | 2
beta-weight
  Frontal Pole (L) | -27.15 (67.37)
  Frontal Orbital Cortex (L) | -88.87 (0.34)
  Superior Frontal Gyrus (R) | -77.23 (68.22)

3. Secondary Outcome: Changes in Endothelial Function at 6 Months
Description: Changes in endothelial function will be measured using brachial artery flow-mediated dilation at baseline, 6 months
Time Frame: Baseline, 6 months
Population: This outcome cannot be reported due to corruption of the collected image data.
Arm/Group | Placebo | GnRH Agonist
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Changes in Endothelial Function at 9 Months
Description: Changes in endothelial function will be measured using brachial artery flow-mediated dilation at baseline, 9 months
Time Frame: Baseline, 9 months
Population: Outcome measure was collected for a subset of the GnRH agonist arm only. This outcome cannot be reported due to corruption of the collected image data.
Arm/Group | GnRH Agonist
Number analyzed (Participants) | 0

5. Secondary Outcome: Changes in Artery Compliance at 6 Months
Description: Changes in carotid artery compliance will be measured using ultrasound in at baseline, 6 months.
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: mm^2/mmhgx10^-1
Arm/Group | Placebo | GnRH Agonist
Number analyzed (Participants) | 4 | 3
mm^2/mmhgx10^-1 | -0.048 (0.057) | -0.095 (0.011)

6. Secondary Outcome: Changes in Artery Compliance at 9 Months
Description: Changes in carotid artery compliance will be measured using ultrasound in at baseline, 9 months.
Time Frame: Baseline, 9 months
Population: Outcome measure was only collected for a subset of the GnRH agonist arm.
Measure: Mean (Standard Deviation); unit: mm^2/mmhgx10^-1
Arm/Group | GnRH Agonist
Number analyzed (Participants) | 2
mm^2/mmhgx10^-1 | -0.002 (0.006)

7. Secondary Outcome: Changes in Executive Cognitive Function: Trails A, 6 Months
Description: Change in time (seconds) to complete Trails A test between baseline and 6 months. Negative value indicates faster time (better performance) at 6 months compared to baseline.
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Placebo | GnRH Agonist
Number analyzed (Participants) | 3 | 8
seconds | 2.79 (8.54) | -5.82 (3.11)

8. Secondary Outcome: Changes in Executive Cognitive Function: Trails A, 9 Months
Description: Change in time (seconds) to complete Trails A test between baseline and 9 months. Negative value indicates faster time (better performance) at 9 months compared to baseline.
Time Frame: Baseline, 9 months
Population: Outcome measure was only collected for a subset of the GnRH agonist arm.
Measure: Mean (Standard Deviation); unit: time (seconds)
Arm/Group | GnRH Agonist
Number analyzed (Participants) | 3
time (seconds) | -5.46 (7.12)

9. Secondary Outcome: Changes in Executive Cognitive Function: RAVLT, 6 Months
Description: Change in Rey Auditory Verbal Learning Test from baseline to 6 months.
  Score is the change in the number of items correct on delayed recall trial. Scores on the RAVLT range from 0-15 with higher scores indicating better performance. A positive change indicates improvement in recall.
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: number of items recalled
Arm/Group | Placebo | GnRH Agonist
Number analyzed (Participants) | 3 | 8
number of items recalled | -1.00 (2.65) | -1.38 (1.85)

10. Secondary Outcome: Changes in Executive Cognitive Function: RAVLT, 9 Months
Description: Change in Rey Auditory Verbal Learning Test from baseline to 9 months.
  Score is the change in the number of items correct on delayed recall trial. Scores on the RAVLT range from 0-15 with higher scores indicating better performance. A positive change indicates improvement in recall.
Time Frame: Baseline, 9 months
Population: Outcome measure was only collected for a subset of the GnRH agonist arm.
Measure: Mean (Standard Deviation); unit: number of items recalled
Arm/Group | GnRH Agonist
Number analyzed (Participants) | 3
number of items recalled | 0 (2.00)

11. Secondary Outcome: Changes in Executive Cognitive Function: Trails B, 6 Months
Description: Change in time (seconds) to complete Trails B test between baseline and 6 months. Negative value indicates faster time (better performance) at 6 months compared to baseline.
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: time (seconds)
Arm/Group | Placebo | GnRH Agonist
Number analyzed (Participants) | 3 | 8
time (seconds) | 14.23 (4.77) | -4.32 (16.27)

12. Secondary Outcome: Changes in Executive Cognitive Function: Trails B, 9 Months
Description: Change in time (seconds) to complete Trails B test between baseline and 9 months. Negative value indicates faster time (better performance) at 9 months compared to baseline.
Time Frame: Baseline, 9 months
Population: Outcome measure was only collected for a subset of the GnRH agonist arm.
Measure: Mean (Standard Deviation); unit: time (seconds)
Arm/Group | GnRH Agonist
Number analyzed (Participants) | 3
time (seconds) | 14.14 (12.09)

13. Secondary Outcome: Changes in Executive Cognitive Function: Stroop, 6 Months
Description: Change in number of correct responses in one minute on Stroop Color Word Interference test between baseline and 6 months. A positive number indicates more items correct indicating better performance. There is no maximum score because the test measures how many correct responses a participant can return within one minute (minimum = 0), however 40 or fewer is considered low. The change in the number of correct responses is reported, and so a positive number indicates more correct responses and better/improved cognitive function.
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: number correct in one minute
Arm/Group | Placebo | GnRH Agonist
Number analyzed (Participants) | 3 | 8
number correct in one minute | -0.67 (10.97) | 0.25 (13.76)

14. Secondary Outcome: Changes in Executive Cognitive Function: Stroop, 9 Months
Description: Change in number of correct responses in one minute on Stroop Color Word Interference test between baseline and 9 months. Positive number indicates more items correct indicating better performance. There is no maximum score because the test measures how many correct responses a participant can return within one minute (minimum = 0), however 40 or fewer is considered low. The change in the number of correct responses is reported, and so a positive number indicates more correct responses and better/improved cognitive function.
Time Frame: Baseline, 9 months
Population: Outcome measure was only collected for a subset of the GnRH agonist arm.
Measure: Mean (Standard Deviation); unit: number correct in one minute
Arm/Group | GnRH Agonist
Number analyzed (Participants) | 3
number correct in one minute | 7.33 (3.06)

15. Secondary Outcome: Changes in Executive Cognitive Function: Digits Span Forward and Backward, 6 Months
Description: Change in score on the Digit Span Test between baseline and 6 month. Raw scores on the Digit Span test range from 0-16 (Digits Forward) and 0-10 (Digits Backward) with higher scores indicating better performance. A positive change score indicates improved performance.
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: number of correct trials
Arm/Group | Placebo | GnRH Agonist
Number analyzed (Participants) | 3 | 8
number of correct trials
  Digits Forward (trials correct) | 1.00 (1.00) | -0.88 (1.89)
  Digits Backward (trials correct) | -0.67 (3.06) | 0.00 (1.51)

16. Secondary Outcome: Changes in Executive Cognitive Function: Digits, 9 Months
Description: Change in score on the Digit Span Test between baseline and 9 months. Raw scores on the Digit Span test range from 0-16 (Digits Forward) and 0-10 (Digits Backward) with higher scores indicating better performance. A positive change score indicates improved performance.
Time Frame: Baseline, 9 months
Population: Outcome measure was only collected for a subset of the GnRH agonist arm.
Measure: Mean (Standard Deviation); unit: number of trials correct
Arm/Group | GnRH Agonist
Number analyzed (Participants) | 3
number of trials correct
  Digits Forward (trials correct) | 1.00 (3.61)
  Digits Backward (trials correct) | 1.0 (1.0)

17. Secondary Outcome: Changes in Executive Cognitive Function: Controlled Oral Word Association Test, 6 Months
Description: Change in sum of scores on 3 COWAT trials (letters, F, A, and S) between baseline and 6 months. Participants are given one minute to think up as many words as they can associated with each letter (F, A, or S). Raw scores are the total number of words generated across all trials. Higher scores indicate more words generated and better performance. Positive change score indicates an increase in words generated, or improved performance.
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: words generated
Arm/Group | Placebo | GnRH Agonist
Number analyzed (Participants) | 3 | 8
words generated | -5.33 (7.77) | 0.25 (9.50)

18. Secondary Outcome: Changes in Executive Cognitive Function: Controlled Oral Word Association Test, 9 Months
Description: Change in sum of scores on 3 COWAT trials (letters, F, A, and S) between baseline and 9 months. Participants are given one minute to think up as many words as they can associated with each letter (F, A, or S). Raw scores are the total number of words generated across all trials. Higher scores indicate more words generated and better performance. Positive change score indicates an increase in words generated, or improved performance.
Time Frame: Baseline, 9 months
Measure: Mean (Standard Deviation); unit: words generated
Arm/Group | GnRH Agonist
Number analyzed (Participants) | 3
words generated | 7.33 (5.51)

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Placebo | GnRH Agonist
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/12
Other Adverse Events (participants affected / at risk) | 0/5 | 1/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=5) | GnRH Agonist (N=12)
calcification of the falx cerebri right of midline (Nervous system disorders) | 0 (0) | 1 (1) — Incidental finding on MRI: There is a prominent (T1/T2 hypo intense) calcification of the falx cerebri right of midline at the level of the precentral gyrus. This is an incidental finding of no clinical importance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-12): https://cdn.clinicaltrials.gov/large-docs/98/NCT02122198/Prot_SAP_000.pdf